CLINICAL TRIAL: NCT03257280
Title: Impact on the Hospital Stay, of an Early Oral Nutrition Protocol Applied to Gastric Cancer Patients After Total Gastrectomy: A Prospective Randomized Control Trial (DOPGT_2015)
Brief Title: Trial on Impact on the Hospital Stay, of an Early Oral Nutrition Protocol Applied to Patients After Total Gastrectomy. (DOPGT_2015)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Leandre Farran Teixidor, Chief of oesophagogastric surgery department, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DOPGT_2015
Record Dates: First submitted 2017-07-07; First posted 2017-08-22 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Early Oral Nutrition After Total Gastrectomy; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early oral nutrition (Experimental): An early oral nutrition with supplements and increased progressively according to an established schedule, start 48 hours after total gastrectomy.
  Interventions: Other: Early oral nutrition
- control group (No Intervention): In our center, the classical postoperative management consisted in one week period of non oral intake and total parenteral nutrition. At the 7 day, an oral contrast image is performed to prove the correct function of the anastomosis, in witch case, a three days progressive oral diet is begin.

INTERVENTIONS:
Other: Early oral nutrition — An early oral nutrition with supplements and increased progressively according to an established schedule, start 48 hours after total gastrectomy.
  Arms: Early oral nutrition

SUMMARY:
This is a prospective randomized controlled clinical trial to clarify the effect of early oral nutrition introduction after total gastrectomy in gastric cancer patients on the length of hospital stay, comparing an experimental group vs control group.

DETAILED DESCRIPTION:
The total gastrectomy is a high complexity surgery that involves a high morbid-mortality. In our center, the postoperative management consisted in 1 week period of non oral intake and total parenteral nutrition. At the 7 day, an oral contrast image is performed to prove the correct function of the anastomosis, in witch case, a progressive oral diet is begin.

In the late 90s, the Fast-track concept (or multimodal perioperative patient care) was introduced in the surgical patients attempting to improve their postoperative course. This new concept includes the preoperative advices related to the surgery, the intensive mobilization after surgery, the early oral diet, and to avoid the routinary use of the nasogastric tube. Some groups have been trying to apply this Fast-track program sporadically in patients submitted to an elective total gastrectomy for gastric cancer, even do, there is still no good evidence to sport these practice.

Based on the reasons exposed before, the investigators design a prospective randomized controlled trial in gastric cancer patients underwent on a total gastrectomy comparing two groups. 24 hours after gastrectomy the investigators will administer oral methylene blue and if no evidence of drainage leakage the participants will be randomized into two groups: one of them with our classical postoperative management, and the other one implements an early oral nutrition protocol, having in considerations its effectiveness, security, and impact on the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring radical total gastrectomy for gastric cancer.
* 18 or above years old.
* Acceptance and signing the full informed consent.

Exclusion Criteria:

* Patient with poorly controlled diabetes mellitus (glycosylated hemoglobin levels greater than 7%)
* Emergency surgery.
* Total gastrectomy with esophagus-jejunal manual suture.
* Early dehiscence of esophagus-jejunal anastomosis (first 24 hours).
* Reintervention for abdominal complication in the first 24 hours.
* Surgery involving large intestinal or colon resections.
* Proximal resection margin affected requiring a esophagectomy and reconstruction with coloplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Hospital stay | postoperative 1 day to discharge, up to 1 month after surgery
  Postoperatory hospital stay in days

SECONDARY OUTCOMES:
Mortality | During the admission, two weeks and one month after surgery
  Postoperative Mortality: Deaths occurring during admission and / or within 30 days after surgery or during surgical admission if it lasts longer than 30 days.
Hospital readmissions | Two weeks and one month after surgery
  It will be considered the income produced within 30 days after the surgical intervention in which the cause of the admission is attributed to a complication in relation to the surgical intervention.
Weight | First day of hospital admission, two weeks and one month after surgery
  weight shall be measured in kilograms
Anastomotic dehiscence | postoperative 1 day to discharge, up to 1 month after surgery
  Anastomotic dehiscence: If the intra-abdominal drainage presents a purulent appearance or an amylase determination> 30, suspicion of anastomosis dehiscence will be made; In this situation, a clinical test (intake of methylene blue) radiological test (with oral contrast) or endoscopy will be requested to confirm the diagnosis. Anastomosis dehiscence will be confirmed if any of the following occurs:
  * Exit of methylene blue through intra-abdominal drainage
  * Contrast leakage in a radiological test performed for sepsis
  * Evidence of dehiscence in a fibrogastroscopy
  * Evidence of anastomotic dehiscence during a reintervention
Duodenal stump leak | postoperative 1 day to discharge, up to 1 month after surgery
  Intra-abdominal drainage presents a purulent appearance with amylase determination> 30 and a bilirubin value higher than plasmatic bilirubin.
Paralytic ileus | postoperative 1 day to discharge, up to 1 month after surgery
  When three of the following criteria are met.
  Oral intolerance after the fourth postoperative day Abdominal distention and tympanism No bowel motions or flatus Compatible abdominal x-ray
Intra-Abdominal abscesses | postoperative 1 day to discharge, up to 1 month after surgery
  1. Radiological criteria:
     Air inside the collection Collection with heterogeneous and irregular pickup or wall pickup Collection with heterogeneous content
  2. Isolation of one or more microorganisms in culture after percutaneous collection
Postoperative Hemoperitoneum | postoperative 1 day to discharge, up to 1 month after surgery
  Presence of blood in the abdominal cavity after gastrectomy that needs any kind of treatments
Evisceration | postoperative 1 day to discharge, up to 1 month after surgery
  Extrusion of viscera outside the body through a surgical incision
Superficial Incisional Surgical Site Infection | postoperative 1 day to discharge, up to 1 month after surgery
  Superficial Incisional Surgical Site Infection
  Infection within 30 days after the operation and only involves skin and subcutaneous tissue of the incision and at least one of the following:
  Purulent drainage with or without laboratory confirmation, from the superficial incision.
  Organisms isolated from an aseptically obtained culture of fluid or tissue from the superficial incision.
  At least one of the following signs or symptoms of infection: pain or tenderness, localised swelling, redness, or heat and superficial incision is deliberately opened by surgeon, unless incision is culture-negative.
  Diagnosis of superficial incisional surgical site infection made by a surgeon or attending physician.
Height | First day of hospital admission, two weeks and one month after surgery
  Height shall be measured in meters
Percentage of weight lost | First day of hospital admission, two weeks and one month after surgery
  Percentage of weight lost shall be measured in percentage
Impedancemetry | First day of hospital admission, two weeks and one month after surgery
  The impedanciometry will record:
  Phase-angle Na / K ratio Basal metabolism (Kcal) Fat mass percentage Muscle mass percentage Cell mass percentage Extracellular mass percentage

CONTACTS AND LOCATIONS:
Overall Officials: Leandre Farran Teixidor, PhD, MD, Principal Investigator — Bellvitge University Hospital
Locations (1):
- Leandre Farran Teixidor, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Gonzalez CA, Agudo A. Carcinogenesis, prevention and early detection of gastric cancer: where we are and where we should go. Int J Cancer. 2012 Feb 15;130(4):745-53. doi: 10.1002/ijc.26430. Epub 2011 Oct 20. PMID 21918974
- [Background] Allum WH, Blazeby JM, Griffin SM, Cunningham D, Jankowski JA, Wong R; Association of Upper Gastrointestinal Surgeons of Great Britain and Ireland, the British Society of Gastroenterology and the British Association of Surgical Oncology. Guidelines for the management of oesophageal and gastric cancer. Gut. 2011 Nov;60(11):1449-72. doi: 10.1136/gut.2010.228254. Epub 2011 Jun 24. No abstract available. PMID 21705456
- [Background] Van Cutsem E, Dicato M, Geva R, Arber N, Bang Y, Benson A, Cervantes A, Diaz-Rubio E, Ducreux M, Glynne-Jones R, Grothey A, Haller D, Haustermans K, Kerr D, Nordlinger B, Marshall J, Minsky BD, Kang YK, Labianca R, Lordick F, Ohtsu A, Pavlidis N, Roth A, Rougier P, Schmoll HJ, Sobrero A, Tabernero J, Van de Velde C, Zalcberg J. The diagnosis and management of gastric cancer: expert discussion and recommendations from the 12th ESMO/World Congress on Gastrointestinal Cancer, Barcelona, 2010. Ann Oncol. 2011 Jun;22 Suppl 5:v1-9. doi: 10.1093/annonc/mdr284. PMID 21633049
- [Background] Viudez-Berral A, Miranda-Murua C, Arias-de-la-Vega F, Hernandez-Garcia I, Artajona-Rosino A, Diaz-de-Liano A, Vera-Garcia R. Current management of gastric cancer. Rev Esp Enferm Dig. 2012 Mar;104(3):134-41. doi: 10.4321/s1130-01082012000300006. PMID 22449155
- [Background] Okines A, Verheij M, Allum W, Cunningham D, Cervantes A; ESMO Guidelines Working Group. Gastric cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2010 May;21 Suppl 5:v50-4. doi: 10.1093/annonc/mdq164. No abstract available. PMID 20555102
- [Background] Wong J, Kelly KJ, Mittra A, Gonen M, Allen P, Fong Y, Coit D. Rt-PCR increases detection of submicroscopic peritoneal metastases in gastric cancer and has prognostic significance. J Gastrointest Surg. 2012 May;16(5):889-96; discussion 896. doi: 10.1007/s11605-012-1845-2. Epub 2012 Feb 24. PMID 22362071
- [Background] Takata A, Kurokawa Y, Fujiwara Y, Nakamura Y, Takahashi T, Yamasaki M, Miyata H, Nakajima K, Takiguchi S, Mori M, Doki Y. Prognostic value of CEA and CK20 mRNA in the peritoneal lavage fluid of patients undergoing curative surgery for gastric cancer. World J Surg. 2014 May;38(5):1107-11. doi: 10.1007/s00268-013-2385-y. PMID 24305936
- [Background] Washington K. 7th edition of the AJCC cancer staging manual: stomach. Ann Surg Oncol. 2010 Dec;17(12):3077-9. doi: 10.1245/s10434-010-1362-z. No abstract available. PMID 20882416
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2010 (ver. 3). Gastric Cancer. 2011 Jun;14(2):113-23. doi: 10.1007/s10120-011-0042-4. No abstract available. PMID 21573742
- [Background] Feng F, Ji G, Li JP, Li XH, Shi H, Zhao ZW, Wu GS, Liu XN, Zhao QC. Fast-track surgery could improve postoperative recovery in radical total gastrectomy patients. World J Gastroenterol. 2013 Jun 21;19(23):3642-8. doi: 10.3748/wjg.v19.i23.3642. PMID 23801867
- [Background] Deguchi Y, Fukagawa T, Morita S, Ohashi M, Saka M, Katai H. Identification of risk factors for esophagojejunal anastomotic leakage after gastric surgery. World J Surg. 2012 Jul;36(7):1617-22. doi: 10.1007/s00268-012-1559-3. PMID 22415758
- [Background] Schietroma M, Cecilia EM, Carlei F, Sista F, De Santis G, Piccione F, Amicucci G. Prevention of anastomotic leakage after total gastrectomy with perioperative supplemental oxygen administration: a prospective randomized, double-blind, controlled, single-center trial. Ann Surg Oncol. 2013 May;20(5):1584-90. doi: 10.1245/s10434-012-2714-7. Epub 2012 Oct 26. PMID 23099730
- [Background] Kucukay F, Okten RS, Parlak E, Disibeyaz S, Ozogul Y, Bostanci EB, Olcer T. Self-expanding covered metallic stent treatment of esophagojejunostomy fistulas. Abdom Imaging. 2013 Apr;38(2):244-8. doi: 10.1007/s00261-012-9895-1. PMID 22527158
- [Background] Lang H, Piso P, Stukenborg C, Raab R, Jahne J. Management and results of proximal anastomotic leaks in a series of 1114 total gastrectomies for gastric carcinoma. Eur J Surg Oncol. 2000 Mar;26(2):168-71. doi: 10.1053/ejso.1999.0764. PMID 10744938
- [Background] Langer FB, Wenzl E, Prager G, Salat A, Miholic J, Mang T, Zacherl J. Management of postoperative esophageal leaks with the Polyflex self-expanding covered plastic stent. Ann Thorac Surg. 2005 Feb;79(2):398-403; discussion 404. doi: 10.1016/j.athoracsur.2004.07.006. PMID 15680802
- [Background] Bardram L, Funch-Jensen P, Jensen P, Crawford ME, Kehlet H. Recovery after laparoscopic colonic surgery with epidural analgesia, and early oral nutrition and mobilisation. Lancet. 1995 Mar 25;345(8952):763-4. doi: 10.1016/s0140-6736(95)90643-6. PMID 7891489
- [Background] Wilmore DW, Kehlet H. Management of patients in fast track surgery. BMJ. 2001 Feb 24;322(7284):473-6. doi: 10.1136/bmj.322.7284.473. No abstract available. PMID 11222424
- [Background] Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. doi: 10.1016/s0002-9610(02)00866-8. PMID 12095591
- [Background] Kehlet H. Future perspectives and research initiatives in fast-track surgery. Langenbecks Arch Surg. 2006 Sep;391(5):495-8. doi: 10.1007/s00423-006-0087-8. Epub 2006 Aug 19. PMID 16924532
- [Background] Kehlet H, Wilmore DW. Evidence-based surgical care and the evolution of fast-track surgery. Ann Surg. 2008 Aug;248(2):189-98. doi: 10.1097/SLA.0b013e31817f2c1a. PMID 18650627
- [Background] Wind J, Polle SW, Fung Kon Jin PH, Dejong CH, von Meyenfeldt MF, Ubbink DT, Gouma DJ, Bemelman WA; Laparoscopy and/or Fast Track Multimodal Management Versus Standard Care (LAFA) Study Group; Enhanced Recovery after Surgery (ERAS) Group. Systematic review of enhanced recovery programmes in colonic surgery. Br J Surg. 2006 Jul;93(7):800-9. doi: 10.1002/bjs.5384. PMID 16775831
- [Background] Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O, Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clin Nutr. 2010 Aug;29(4):434-40. doi: 10.1016/j.clnu.2010.01.004. Epub 2010 Jan 29. PMID 20116145
- [Background] Kehlet H, Slim K. The future of fast-track surgery. Br J Surg. 2012 Aug;99(8):1025-6. doi: 10.1002/bjs.8832. Epub 2012 Jun 14. No abstract available. PMID 22696149
- [Background] Olsen MF, Wennberg E. Fast-track concepts in major open upper abdominal and thoracoabdominal surgery: a review. World J Surg. 2011 Dec;35(12):2586-93. doi: 10.1007/s00268-011-1241-1. PMID 21882022
- [Background] Lassen K, Kjaeve J, Fetveit T, Trano G, Sigurdsson HK, Horn A, Revhaug A. Allowing normal food at will after major upper gastrointestinal surgery does not increase morbidity: a randomized multicenter trial. Ann Surg. 2008 May;247(5):721-9. doi: 10.1097/SLA.0b013e31815cca68. PMID 18438106
- [Background] Hur H, Si Y, Kang WK, Kim W, Jeon HM. Effects of early oral feeding on surgical outcomes and recovery after curative surgery for gastric cancer: pilot study results. World J Surg. 2009 Jul;33(7):1454-8. doi: 10.1007/s00268-009-0009-3. PMID 19399550
- [Background] Lewis SJ, Andersen HK, Thomas S. Early enteral nutrition within 24 h of intestinal surgery versus later commencement of feeding: a systematic review and meta-analysis. J Gastrointest Surg. 2009 Mar;13(3):569-75. doi: 10.1007/s11605-008-0592-x. Epub 2008 Jul 16. PMID 18629592
- [Background] Liu XX, Jiang ZW, Wang ZM, Li JS. Multimodal optimization of surgical care shows beneficial outcome in gastrectomy surgery. JPEN J Parenter Enteral Nutr. 2010 May-Jun;34(3):313-21. doi: 10.1177/0148607110362583. PMID 20467014
- [Background] Wang D, Kong Y, Zhong B, Zhou X, Zhou Y. Fast-track surgery improves postoperative recovery in patients with gastric cancer: a randomized comparison with conventional postoperative care. J Gastrointest Surg. 2010 Apr;14(4):620-7. doi: 10.1007/s11605-009-1139-5. Epub 2010 Jan 28. PMID 20108171
- [Background] Chen Hu J, Xin Jiang L, Cai L, Tao Zheng H, Yuan Hu S, Bing Chen H, Chang Wu G, Fei Zhang Y, Chuan Lv Z. Preliminary experience of fast-track surgery combined with laparoscopy-assisted radical distal gastrectomy for gastric cancer. J Gastrointest Surg. 2012 Oct;16(10):1830-9. doi: 10.1007/s11605-012-1969-4. Epub 2012 Aug 2. PMID 22854954
- [Background] Kim JW, Kim WS, Cheong JH, Hyung WJ, Choi SH, Noh SH. Safety and efficacy of fast-track surgery in laparoscopic distal gastrectomy for gastric cancer: a randomized clinical trial. World J Surg. 2012 Dec;36(12):2879-87. doi: 10.1007/s00268-012-1741-7. PMID 22941233
- [Background] Fujitani K, Tsujinaka T, Fujita J, Miyashiro I, Imamura H, Kimura Y, Kobayashi K, Kurokawa Y, Shimokawa T, Furukawa H; Osaka Gastrointestinal Cancer Chemotherapy Study Group. Prospective randomized trial of preoperative enteral immunonutrition followed by elective total gastrectomy for gastric cancer. Br J Surg. 2012 May;99(5):621-9. doi: 10.1002/bjs.8706. Epub 2012 Feb 24. PMID 22367794
- [Background] Marano L, Porfidia R, Pezzella M, Grassia M, Petrillo M, Esposito G, Braccio B, Gallo P, Boccardi V, Cosenza A, Izzo G, Di Martino N. Clinical and immunological impact of early postoperative enteral immunonutrition after total gastrectomy in gastric cancer patients: a prospective randomized study. Ann Surg Oncol. 2013 Nov;20(12):3912-8. doi: 10.1245/s10434-013-3088-1. Epub 2013 Jul 10. PMID 23838912
- [Background] Braga M, Gianotti L, Vignali A, Di Carlo V. Immunonutrition in gastric cancer surgical patients. Nutrition. 1998 Nov-Dec;14(11-12):831-5. doi: 10.1016/s0899-9007(98)00103-8. PMID 9834924
- [Background] Mabvuure NT, Roman A, Khan OA. Enteral immunonutrition versus standard enteral nutrition for patients undergoing oesophagogastric resection for cancer. Int J Surg. 2013;11(2):122-7. doi: 10.1016/j.ijsu.2012.12.012. Epub 2012 Dec 26. PMID 23274278
- [Background] Mortensen K, Nilsson M, Slim K, Schafer M, Mariette C, Braga M, Carli F, Demartines N, Griffin SM, Lassen K; Enhanced Recovery After Surgery (ERAS(R)) Group. Consensus guidelines for enhanced recovery after gastrectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Br J Surg. 2014 Sep;101(10):1209-29. doi: 10.1002/bjs.9582. Epub 2014 Jul 21. PMID 25047143